CLINICAL TRIAL: NCT01594840
Title: Changing Chat: Diaper Tips to Improve Language Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Dimitri Christakis, Director, Center for Child Health, Behavior, and Development, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Changing chat
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Infants
Keywords: language development; parental interaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Changing chat (Experimental): Diapers will have tips on them
  Interventions: Device: Changing chat
- Control (Active Comparator): Normal diapers
  Interventions: Device: Changing chat

INTERVENTIONS:
Device: Changing chat — Diapers with tips

SUMMARY:
This randomized trial has two sets of diapers-- a normal one and one that has tips for how to talk to and engage your toddler. The investigators are hoping that the intervention improves language development.

ELIGIBILITY:
Inclusion Criteria:

16-18 months of age developmentally normal English speaking

Exclusion Criteria:

-

Ages: 16 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Language development as measured by the Mcarthur Bates CDI | 6 months after

CONTACTS AND LOCATIONS:
Locations (1):
- Odessa Brown, Seattle, Washington, United States